CLINICAL TRIAL: NCT01306201
Title: A Novel Cardio-Respiratory Parameter in a Hospital Setting
Brief Title: Novel Non-Invasive Monitoring Parameter in a Hospital Setting
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0131
Record Dates: First submitted 2011-02-10; First posted 2011-03-01 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
Keywords: Hospital Setting
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-patient Volunteers: In-patients from the hospital who choose to participate in the study

SUMMARY:
Data collected from this study will be used to evaluate the performance of a monitoring algorithm.

DETAILED DESCRIPTION:
The goal of this study is to assess equivalency, performance, and accuracy of a new monitoring algorithm in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years old or older
2. Written informed consent from the patient or their legally authorized representative before initiation of any study-related procedures
3. Subjects on general care floor

Exclusion Criteria:

1. Severe contact allergies to standard adhesive materials
2. Abnormalities that may prevent proper application of the device
3. Women who are pregnant or lactating
4. Subjects with significant arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Care Floor Patients
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bergese, MD, Principal Investigator — The Ohio State Medical Center, Dept of Anesthesia; Robert McIntyre, MD, Principal Investigator — University of Colorado Denver, School of Medicine dept of Surgery Division of GI, Tumor and Endocrine Surgery
Locations (2):
- United States (2):
  - The University of Colorado Health Sciences Center (UCHSC), Denver, Colorado
  - The Ohio State University Medical Center (OSUMC), Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates were February 10, 2011- to March 4th,2011
Groups:
- Respiration Rate in GCF Patients: In-patients from the hospital general care floor, who choose to participate in the study. Participants were monitored for 30 minute periods to collect respiratory rate information from non-invasive sensors.
Period: Overall Study
Arm/Group | Respiration Rate in GCF Patients
Started | 63
Completed | 53 (Total of 10 subjects were excluded from analysis)
Not Completed | 10
Not completed — Arrhythmia | 4
Not completed — Files could not be processed | 3
Not completed — Files unreadable | 3

BASELINE CHARACTERISTICS:
Arm/Group | In-patient Volunteers
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: The Covidien Nellcor Respiration Rate Software Shall Determine Respiration Rate Measured as Mean and Standard Deviation With Accuracy That is Non-inferior to Predicate Device.
Description: Mean and standard deviations of respiration rates collected from patients in the hospital settings were compared between Covidien Respiration Rate Software, Transthoracic Impedance and End-Tidal Carbon Dioxide Waveforms. Each patient served as its own control.
Time Frame: Participants were monitored for average of 30 minutes
Population: 10 participants were excluded from data analysis due to following reasons: unreadable files,arrhythmia,electronic data files coud not be processed
Measure: Mean (Standard Deviation); unit: BrPM (Breaths Per Minute)
Groups:
- Respiration Rate From Covidien Respiration Rate Software: Respiration rate determined by novel plethysmographic analysis
- Respiration Rate From Endtidal Carbon Dioxide Waveform: Respiration rate determined by manual overscoring of capnography waveforms
- Respiration Rate From Transthoracic Impedance: Respiration Rate derived from Transthoracic Impedance
Arm/Group | Respiration Rate From Covidien Respiration Rate Software | Respiration Rate From Endtidal Carbon Dioxide Waveform | Respiration Rate From Transthoracic Impedance
Number analyzed (Participants) | 53 | 53 | 53
BrPM (Breaths Per Minute) | 15.4 (4.0) | 16.0 (4.6) | 16.8 (4.8)

2. Secondary Outcome: The Covidien Nellcor Respiration Rate Software Shall Calculate Respiration Rate With a Root Mean Square Difference (RMSD) of < 3 Breaths Per Minute Compared With a End-Tidal Carbon Dioxide Waveforms, With 95% Confidence.
Description: The data used for analysis consisted of multiple simultaneous measures of RR_TTI, RR_V1.0 and RR_EtCO2 for each subject. Given N sets of simultaneous RR values for each of P patients, the simultaneous RR values were used to calculate a pair of RMSD values for each subject.
  The two RMSD values, RMSDRR_V1.0_vs_EtCO2, and RMSDTTI_vs_EtCO2, quantify the mean absolute difference in simultaneous estimates of respiratory rate between RR_V1.0 compared with RR_EtCO2 and RR_TTI compared with RR_EtCO2, respectively for the subjects with 95% confidence of mean ± 3.38 BrPM. The Measure type is Number and represents the RMSD of Covidien Nellcor Respiration Rate Software
Time Frame: Participants were monitored on average for 30 minutes
Measure: Number; unit: Breaths Per Minute (BrPM)
Groups:
- Overall Study Population: Covidien Respiration Rate, Transthoracic Impedance and Overscored Endtidal Carbon Dioxide derived respiration rates were recorded on all the volunteers simultaneously.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 53
Breaths Per Minute (BrPM) | 1.60

3. Post Hoc Outcome: Calculate Covidien Respiration Rate Software Accuracy as Mean Error +/- Standard Deviation.
Time Frame: Overall average
Measure: Mean (Standard Deviation); unit: Breaths Per Minute (BrPM)
Arm/Group | In-patient Volunteers
Number analyzed (Participants) | 53
Breaths Per Minute (BrPM) | 0.07 (1.98)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | In-patient Volunteers
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No